CLINICAL TRIAL: NCT00231894
Title: Pioglitazone as a Treatment for Lipid and Glucose Abnormalities In Patients With Schizophrenia Treated With Antipsychotic Medication And Potential Effects on Cognitive Function
Brief Title: Pioglitazone as a Treatment for Lipid and Glucose Abnormalities In Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04T-584 Stanley Foundation; 04T-584 (Other Grant/Funding Number: Stanley Foundation)
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Diabetes; Schizophrenia; Insulin Resistance; Cognitive Impairment
Keywords: atypical antipsychotics; hyperglycemia; triglycerides; HDL; cholesterol; insulin resistance; schizophrenia; verbal memory
MeSH Terms: conditions — Diabetes Mellitus; Schizophrenia; Insulin Resistance; Cognitive Dysfunction; Hyperglycemia | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone and life-style group (Active Comparator): Pioglitazone (30-45 mg/daily) plus life-style diet group
  Interventions: Drug: Pioglitazone; Behavioral: Life style diet group
- Placebo and life style group (Placebo Comparator): Placebo capsules daily plus life-style diet group
  Interventions: Behavioral: Life style diet group; Other: Placebo

INTERVENTIONS:
Drug: Pioglitazone — pioglitazone 30-45 mg/day
  Other Names: Actos
  Arms: Pioglitazone and life-style group
Behavioral: Life style diet group — life style diet education group 1x/week
Other: Placebo — placebo comparator capsules
  Arms: Placebo and life style group

SUMMARY:
This is a study with an approved drug for treating type 2 diabetes, for its effects on treating glucose and lipid abnormalities in patients being treated with first or second-generation antipsychotics, and comparison of effects of this drug with another treatment lifestyle modification. Patients who meet inclusion criteria will be treated with pioglitazone for 12 weeks. They will be evaluated for fasting glucose and lipids, glucose-tolerance tests, and neurocognitive battery and tests of verbal memory at baseline and during treatment with pioglitazone.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of pioglitazone added to weight-lifestyle intervention vs. placebo plus lifestyle intervention on reversing or reducing impaired or abnormal triglycerides, HDL and glucose metabolism in schizophrenics treated with first or second-generation antipsychotics.. Another aim is to examine the effects of impaired glucose metabolism on verbal memory and other cognitive function in schizophrenic patients treated with these medications and the relationship to improvements in impaired glucose metabolism to impairments in cognitive function. Clozapine and olanzapine, and some other first or second-generation antipsychotics effective for treating schizophrenia and bipolar disorders, have been reported to be associated with increased incidence of diabetic type metabolic abnormalities, decreases in insulin sensitivity, and abnormal glucose tolerance tests. This can lead to the development of type 2 diabetes and also abnormal lipid metabolic levels which can lead to atherosclerotic changes and increased risk of cardiovascular disease and other diabetes related complications. Drug treatments which could reduce or correct these diabetic metabolic changes would permit many patients to continue to receive the benefits of these antipsychotic medications with reduced drug-induced comorbidity. Previous research using non-psychotic subjects has shown that diabetes and impaired glucose tolerance are associated with cognitive impairments, especially in verbal memory, and provides a rationale for testing whether corrections of impaired glucose metabolism are associated with cognitive improvements in schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be males or females, 18-70 yrs of age, with a diagnosis of schizophrenia or schizoaffective disorder, and currently being treated with olanzapine or clozapine.
2. Patients will have evidence of:

   1. glucose levels indicating at least impaired fasting glucose: fasting glucose 100 mg/dL or 2 hr glucose tolerance test 140 mg/dL, or current treatment with oral antidiabetic drugs with history of hyperglycemia;
   2. Triglyceride levels > 120 mg/dL and/or HDL levels < 40 mg/dL

Exclusion Criteria:

1. Diabetes mellitus, type 1
2. Recent diabetic ketoacidosis;
3. Patients not currently treated with oral antidiabetic drugs but fasting is glucose 140 mg/dL [WHO criteria] on repeat testing in last three months, or random blood glucose >200 mg/dL plus 2 hr glucose on GTT >200 mg/dL; (these patients may need more immediate treatment with antidiabetic drugs and it is less certain if weight-lifestyle treatment would be effective in treating such high glucose levels);
4. Patients with active liver disease with clinical abnormalities which need current treatment, or liver enzymes (Alt) 3 times upper limit for normal values in chart records in last year, or patients who are recorded as positive for hepatitis C;
5. Congestive heart failure (Class III or IV cardiac status) or history of MI in medical record (because pioglitazone can increase blood volume slightly);
6. Hematocrit greater than 10% below normal (hematocrit may be decreased 2 to 4% due to increased plasma volume);
7. Female patients on current oral contraceptives (because pioglitazone may interfere with effects of some oral contraceptives);
8. Patients taking ketoconazole,
9. Patients who have started on atorvastatin or gemfibrozil in the past 2 months or have had a dose increase in atorvastatin in the last month (since these drugs can also lower triglycerides and raise HDL, recent start of therapy with these drugs could be a confound).
10. Patients are not concomitantly treated with aripiprazole or ziprasidone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Smith, MD PhD, Principal Investigator — NYU School of Medicine & Nathan Kline Institute for Psychiatric Research
Locations (1):
- Nathan Kline Institute for Psychiatric Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith RC et al Pioglitazone as a treatment for glucose and lipid abnormalities in schizophrenic patents: A double-blind placebo controlled trial. NCDEU 51lst Annual Meeting Oral Presentation Abstract Book, 2011, p.13.
- [Result] Smith RC, Jin H, Li C, Bark N, Shekhar A, Dwivedi S, Mortiere C, Lohr J, Hu Q, Davis JM. Effects of pioglitazone on metabolic abnormalities, psychopathology, and cognitive function in schizophrenic patients treated with antipsychotic medication: a randomized double-blind study. Schizophr Res. 2013 Jan;143(1):18-24. doi: 10.1016/j.schres.2012.10.023. Epub 2012 Nov 29. PMID 23200554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at 6 U.S. sites and one site in Shanghai, China
Groups:
- Pioglitazone: Pioglitazone (30-45 mg/daily) plus life-style diet education group
- Placebo: Placebo capsules daily plus life-style diet education group
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 31 | 25
Completed | 30 | 24
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone: pioglitazone
- Placebo: placebo
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 30 | 24 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.06) | 48.5 (10.17) | 47.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 27 | 21 | 48
Region of Enrollment [Number; unit: participants]
  United States | 25 | 19 | 44
  China | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Triglycerides at 3 Months ( 3 Months-baseline) US Sample
Time Frame: pre-treatment and during 3 months of treatment
Population: Data is from participants at U.S. sites N=44, Pioglitazone =25, Placebo =19, who had values of triglycerides at baseline and three months followup. See table 2 of published paper given in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Pioglitazone: pioglitazone and life-style diet group
- Placebo: placebo and life-style diet group
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 25 | 19
mg/dL | -49.65 (24.01) | 30.99 (26.82)

2. Primary Outcome: Change From Baseline in Serum HDL at 3 Months (3 Months-baseline) US Sample
Description: serum high density lipoprotein (HDL)
Time Frame: pre-treatment and during 3 months of treatment
Population: Data is from participants at U.S. sites N=44, Pioglitazone =25, Placebo =19, who had values of HDL at baseline and three months followup. See table 2 of published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Piogltiazone: pioglitazone and life-style diet group
  Pioglitazone: pioglitazone 15-45 mg/day
  Life style diet group: life style diet education group 1x/week
- Placebo: placebo and life-style diet group
  Life style diet group: life style diet education group 1x/week
  placebo: placebo comparator
Arm/Group | Piogltiazone | Placebo
Number analyzed (Participants) | 25 | 19
mg/dL | 4.62 (1.77) | -2.59 (2.11)

3. Primary Outcome: Change From Baseline in Serum Glucose at 3 Months (3 Months-baseline) US Sample
Time Frame: pretreatment and during 3 months of drug treatment
Population: Data is from participants at U.S. sites N=44, Pioglitazone =25, Placebo =19, who had values of serum glucose at baseline and three months follow-up. See table 2 of published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 25 | 19
mg/dL | 0.02 (8.14) | 24.20 (8.63)

4. Primary Outcome: 2 Hour Glucose From Glucose Tolerance Test US Sample
Description: difference between 2 hr glucose for GTT test at baseline vs after 3 months of drug treatment
Time Frame: between baseline and 3 months of study drug treatment
Population: Data is from participants at U.S. sites N=44, Pioglitazone =25, Placebo =19, who had values of serum glucose at 2-hour point in glucose tolerance test at baseline and three months follow-up. See table 2 of published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 25 | 19
mg/dL | -24.19 (17.03) | 15.19 (17.75)

5. Secondary Outcome: Change in RBANS List Recognition Scores at 3 Months (3 Months-baseline) US Sample
Description: The scale is Repeatable Battery for the Assessment to Neuropsychological Status (RBANS). This scale measure cognitive function in patients with schizophrenia. Range for list learning sub-score is 0 to 20 . Higher values indicate better performance. For change score (3 months -baseline) positive values indicate improved performance for this cognitive function and negative values indicate poorer performance on this cognitive function.
Time Frame: pre-treatment and 3 months of treatment
Population: Data is from participants at U.S. sites N=43, Pioglitazone =25, Placebo =18, who had scores of RBANS List learning at 2-hour point at baseline and three months follow-up. See table 2 of published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: Units on RBANS scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 25 | 19
Units on RBANS scale | 0.27 (0.41) | -1.11 (0.44)

6. Secondary Outcome: Change From Baseline in Serum Glucose at 3 Months ( 3 Months -Baseline) China Sample
Time Frame: pretreatment and during 3 months of drug treatment
Population: Data is from participants at China site N=10, Pioglitazone =5, Placebo =5, who had values of fasting glucose at baseline and three months follow-up. See published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 5
mg/dL | -13.33 (11.08) | -11.5 (3.44)

7. Secondary Outcome: Change From Baseline in Serum Triglycerides at 3 Months (3 Months-baseline) China Sample
Time Frame: pretreatment and during 3 months of drug treatment
Population: Data is from participants at China site N=10, Pioglitazone =5, Placebo =5, who had values of triglycerides at baseline and three months followup. See published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 5
mg/dL | 32.56 (24.76) | -79.12 (40.72)

8. Secondary Outcome: 2 Hour Glucose From Glucose Tolerance Test China Sample
Description: difference between 2 hr glucose for GTT test at baseline vs after 3 months of drug treatment
Time Frame: between baseline and 3 months of study drug treatment
Population: Data is from participants at china site N=10, Pioglitazone =5, Placebo =5, who had values of serum glucose at 2-hour point in glucose tolerance test at baseline and three months follow-up. See published paper and its supplementary data paper cited in reference for further details.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 5
mg/dL | -6.82 (21.28) | -40.72 (21.28)

9. Secondary Outcome: Change From Baseline in Serum HDL at 3 Months (3 Months-baseline) China Site
Time Frame: pretreatment and during 3 months of drug treatment
Population: Data is from participants at china. site N=10, Pioglitazone =5, Placebo =5, who had values of HDL at baseline and three months followup. See of published paper and its supplementary data paper cited in reference for further details
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 5
mg/dL | 6.52 (1.14) | 7.72 (3.37)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/25
Other Adverse Events (participants affected / at risk) | 1/31 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=31) | Placebo (N=25)
glucose increase (Endocrine disorders) | 0 (0) | 1 (1) — One subject had very high glucose values (376 fasting; 530 hour one GTT). It was determined the patient was on a placebo. There was a gap in the patient's insulin coverage..
glucose increase (Endocrine disorders) | 0 (0) | 1 (1) — Patient had high glucose levels and was determined to be on placebo arm of study.
high CPK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Increased in CPK which was not attributable to the study medication (pioglitazone or placebo), but to another medication that the patient was on (gemfibrozil) which the patient had been prescribed previously by this clinical physician..

LIMITATIONS AND CAVEATS:
Sufficient RBANS data at baseline and 3 months followup for China sample was not available for analysis. Subjects failed to complete scales or complete scales with sufficient data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No